CLINICAL TRIAL: NCT06448988
Title: Evaluation of Respiratory Mechanics in Supine and PARK-bench Positions in Patients Undergoing Elective Neurosurgery: a Cross-over Physiological Study
Brief Title: Evaluation of Respiratory Mechanics in Supine and PARK-bench Positions (SPARK)
Acronym: SPARK
Status: Enrolling by invitation | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: FPG ID 6738
Record Dates: First submitted 2024-05-28; First posted 2024-06-07 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Ventilation Therapy; Complications; Ventilator-Induced Lung Injury
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Supine position: To evaluate, during the procedure, the variation in regional distribution of intrapulmonary volume in the dependent and non-dependent lung regions in patients undergoing neurosurgical intervention between supine and Park-Bench position.
  Interventions: Other: Park Bench position

INTERVENTIONS:
Other: Park Bench position — To evaluate, during the procedure, the variation in regional distribution of intrapulmonary volume in the dependent and non-dependent lung regions in patients undergoing neurosurgical intervention between supine and Park-Bench position.

SUMMARY:
The primary objective of this prospective observational physiological study is to evaluate the variation in regional distribution of intrapulmonary volume in the dependent and non-dependent lung regions in patients undergoing neurosurgical intervention between supine and Park-Bench position.

DETAILED DESCRIPTION:
The Park-Bench position is a variant of the lateral position used in neurosurgical interventions where lesions of the posterior cranial fossa and ponto-cerebellar angle need to be approached. The patient is placed in a lateral-oblique position with the arm on the side they are lying on extending out of the operating bed and supported by an external support. The head is fixed in flexion and rotation with the Mayfield headrest immobilizing the head, allowing exposure of the surgical region of interest.

In the lateral decubitus position, several factors contribute to changing respiratory mechanics: airway resistance increases and compliance decreases.

Furthermore, the gravitational gradient is altered, which is one of the main factors in the regional distribution of intrapulmonary air volume and tidal volume distribution: the phenomenon of overdistension of the non-dependent lung and collapse of the dependent lung could occur.

Fully understanding these physiological changes could optimize mechanical ventilation settings and thus avoid causing damage to lung parenchyma (Ventilator-Induced Lung Injury).

The primary hypothesis of this physiological study is to evaluate changes in regional distribution of intrapulmonary volume when transitioning from the supine position to the Park-Bench position.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Patients scheduled for elective neurosurgery in Park-Bench position.

Exclusion Criteria:

* Age < 18
* BMI > 30 kg/m2
* Obstructive or restrictive lung disease with oxygen supplementation
* Pacemaker
* Pregnancy
* Absence of history of pulmonary embolism, thoracic surgery or chest wall abnormalities, organ transplant, lung metastases
* New York Heart Association >2 or hemodynamic instability (Mean Arterial Pressure<60mHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will enroll all patients scheduled for elective neurosurgery in Park-Bench position in Fondazione Policlinico Universitario "Agostino Gemelli", Rome, Italy
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Variation in tidal volume distribution in the dependent and non-dependent lung during neurosurgical intervention, from supine to Park Bench position. | Variation, during the procedure, in tidal volume distribution in the dependent and non-dependent lung during neurosurgical intervention, from supine to Park Bench position.
  Variation in tidal volume distribution in the dependent and non-dependent lung during neurosurgical intervention, from supine to Park Bench position.

SECONDARY OUTCOMES:
Airway closure incidence in the supine and Park Bench position | Airway closure incidence, during the procedure, in the supine and Park Bench position
  Airway closure incidence in the supine and Park Bench position

CONTACTS AND LOCATIONS:
Overall Officials: Giuliano Ferrone, MD, Principal Investigator — Fondazione Policlinico Gemelli, Rome
Locations (1):
- Fondazione Policlinico Gemelli, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grieco DL, Anzellotti GM, Russo A, Bongiovanni F, Costantini B, D'Indinosante M, Varone F, Cavallaro F, Tortorella L, Polidori L, Romano B, Gallotta V, Dell'Anna AM, Sollazzi L, Scambia G, Conti G, Antonelli M. Airway Closure during Surgical Pneumoperitoneum in Obese Patients. Anesthesiology. 2019 Jul;131(1):58-73. doi: 10.1097/ALN.0000000000002662. PMID 30882475
- [Result] Mezidi M, Guerin C. Effects of patient positioning on respiratory mechanics in mechanically ventilated ICU patients. Ann Transl Med. 2018 Oct;6(19):384. doi: 10.21037/atm.2018.05.50. PMID 30460258